CLINICAL TRIAL: NCT00813475
Title: Clinical Outcome of Tight Glucose Control of Diabetic Patients Hospitalized In General Internal Medicine Wards A National Israeli Study
Brief Title: Effect of Diabetes Control on Outcome in Hospitalized Patients: A National Israeli Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Andreas E. Buchs, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 184-08
Record Dates: First submitted 2008-12-21; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes
Keywords: cardio vascular outcome
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tight control (Experimental)
  Interventions: Drug: Basal bolus insulin regimen (tight glucose control)
- standard control (Experimental): basal bolus insulin regimen
  Interventions: Drug: Basal bolus insulin regimen (standard control)

INTERVENTIONS:
Drug: Basal bolus insulin regimen (tight glucose control) — Basal bolus insulin regimen
  Arms: tight control
Drug: Basal bolus insulin regimen (standard control) — basal bolus insulin regimen
  Arms: standard control

SUMMARY:
To test whether tight glucose control is associated with better clinical outcome compared to less-tight control, among diabetic patients hospitalized in internal medicine wards.

DETAILED DESCRIPTION:
Patient characteristics:

Patients admitted to internal medicine departments in public hospitals of Israel who have pre-admission diagnosis of diabetes, or have a random plasma glucose >200 mg/dl on admission

Eligibility criteria

1. Age: >18 years
2. Fasting plasma glucose > 140 mg/dl or non-fasting plasma glucose >200 mg/dl in two separate blood tests if non-diabetic, or in a single blood test if have pre-diagnosed diabetes
3. Able to understand the study objective and methods and willing to provide a written informed consent
4. No significant liver disease
5. Serum creatinine <2.0 mg/dl

Exclusion criteria

1. Significant cognitive impairment
2. History of hypoglycemia unawareness or clinical autonomic diabetic neuropathy
3. Known allergy to insulin analogues
4. Diabetic ketoacidosis or non-ketotic hyperosmolar coma on admission

Process of patient recruitment and randomization:

1. Enrolment of eligible patients signing the informed consent.
2. Assignment of patients to different treatment arms according to randomization scheme provided by the central organizing committee.
3. The ratio of patients' assignment to the active or to the control study arm will be 1:1 for each participating ward.

Protocol:

Basal bolus insulin treatment will be applied to achieve tight glucose target (mean fasting blood glucose<130 mg/dl and not above 180 mg/dl during the day) compared to patients treated to achieve less tight glucose targets (mean fasting blood glucose<200 mg/dl and not above 220 mg/dl during the day)will influence cardiovascular and general clinical outcome.

Primary outcome: All-cause mortality (including in-hospital and up to 12 months post discharge) or re-admission to hospital

Secondary outcomes:

Total number of in-hospital days during one year follow-up (including the index hospital admission)

The rate of any major clinical events (all-cause mortality, hospital acquired infection, organ failure, need of ventilation support, need of vasoactive amine administration, need of central line insertion, hospital admission for stroke, acute coronary event, severe bacterial or fungal infection) during one year follow-up

Hypoglycemic events during index hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >18 years
2. Fasting plasma glucose > 140 mg/dl or non-fasting plasma glucose >200 mg/dl in two separate blood tests if non-diabetic, or in a single blood test if have pre-diagnosed diabetes
3. Able to understand the study objective and methods and willing to provide a written informed consent
4. No significant liver disease
5. Serum creatinine <2.0 mg/dl

   -

Exclusion Criteria:

1. Significant cognitive impairment
2. History of hypoglycemia unawareness or clinical autonomic diabetic neuropathy
3. Known allergy to insulin analogues
4. Diabetic ketoacidosis or non-ketotic hyperosmolar coma on admission

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality (including in-hospital and up to 12 months post discharge) or re-admission to hospital | 1.5 years

SECONDARY OUTCOMES:
Total # of in-hospital days during 1 year follow-up.The rate of any major clinical events during 1 year follow-up. Hypoglycemic events during index hospital stay | 1.5

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel